CLINICAL TRIAL: NCT07350889
Title: Effects of a Specific Dietary Program on Overweight/Obese Women With Polycystic Ovary Syndrome: A Multicenter, Prospective, Randomized Controlled Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Jinan Central Hospital (Other); Civil Aviation General Hospital (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2025]438-002
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific dietary intervention (Experimental)
  Interventions: Behavioral: Specific dietary intervention group
- Conventional intervention (Active Comparator)
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: Specific dietary intervention group — 1. Energy Levels and Individualized Matching The dietary intervention includes three energy levels: 1200 kcal, 1400 kcal, and 1600 kcal. Based on height, weight, basal metabolic rate, and weight loss goals, participants are matched to the appropriate energy level. The nutrition team will adjust the energy level and dietary plan every 4 weeks based on weight changes and metabolic feedback, with the intervention continuing for 24 weeks.
  2. Nutritional Composition and Base Formula Design The plan consists of 1000 kcal for lunch and dinner daily, with a focus on high protein (>80g) and high fiber (>30g) to support weight management and improve metabolic status. This intervention will continue for 24 weeks.
  3. Food Ingredients and Intervention Frequency The intervention uses natural ingredients, with at least 12 types of foods daily. Participants will have 5 days of standardized meals and 2 free eating days per week to improve adherence. The intervention will last for 24 weeks.
  Arms: Specific dietary intervention
Behavioral: Conventional intervention — The dietary intervention involves a 20% reduction in total caloric intake, with a balanced distribution of nutrients to ensure adequate intake of essential macronutrients and micronutrients. The intervention will be implemented over a period of 24 weeks.
  Arms: Conventional intervention

SUMMARY:
The goal of this clinical trial is to investigate the effects of a specific dietary program on overweight or obese patients with polycystic ovary syndrome (PCOS) through a multicenter, randomized, controlled, prospective study design.

The main questions it aims to answer are:

1. Does the specific dietary program increase the clinical remission rate of PCOS in overweight or obese patients?
2. Does the specific dietary program improve metabolic and anthropometric outcomes in overweight or obese patients with PCOS compared with conventional intervention?

Researchers will compare the effects of a specific dietary program versus conventional intervention on clinical remission rates, metabolic outcomes, and anthropometric measures in overweight or obese patients with PCOS.

Participants will:

1. Receive either a specific dietary intervention or conventional intervention for 24 weeks.
2. Undergo assessments every 12 weeks throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged 18-49 years.
2. Body mass index (BMI) ≥ 24 kg/m² and waist circumference ≥ 85 cm.
3. Diagnosis of polycystic ovary syndrome (PCOS) based on the 2003 Rotterdam consensus, defined by the presence of at least two of the following three criteria: (i) Oligo-ovulation and/or anovulation; (ii) Clinical and/or biochemical signs of hyperandrogenism; (iii) Polycystic ovarian morphology on ultrasonography, defined as the presence of ≥12 follicles measuring 2-9 mm in diameter in each ovary and/or increased ovarian volume ≥10 cm³.
4. Menstrual irregularity.
5. Use of reliable non-hormonal contraception throughout the study period.
6. Provision of written informed consent.

Exclusion Criteria:

1. Participants with non-classical 21-hydroxylase deficiency, hyperprolactinemia, Cushing's disease, or adrenal tumors will be excluded from the study.
2. Participants who are postmenopausal or perimenopausal, as well as those who are pregnant, planning pregnancy, or currently lactating, will be excluded.
3. Participants with a history of substance abuse, acute infectious diseases, or diabetes mellitus will not be eligible for inclusion.
4. Participants with a history of malignancy within the past 5 years or with current malignant disease will be excluded.
5. Participants with a history of gallstones or gout will be excluded from the study.
6. Participants with poorly controlled thyroid disorders, regardless of etiology, will be excluded.
7. Participants who have been diagnosed with an eating disorder within the past 12 months will be excluded.
8. Participants with known intolerance or allergy to components of the study dietary plan, such as soy, lactose, or gluten, or those diagnosed with celiac disease, will be excluded.
9. Participants who have used medications that may affect reproductive or metabolic outcomes within the past 3 months will be excluded, including oral hormonal contraceptives or hormonal implants; anti-androgens (e.g., spironolactone, flutamide, finasteride); metformin or other insulin-sensitizing agents; clomiphene citrate or estrogen modulators; gonadotropin-releasing hormone (GnRH) modulators (e.g., leuprolide); minoxidil; weight-loss medications; or other drugs that may influence appetite, such as oral corticosteroids.
10. Participants with severe hepatic impairment, defined as alanine aminotransferase (ALT) > 100 U/L or aspartate aminotransferase (AST) > 100 U/L, will be excluded.
11. Participants with severe renal impairment, defined as an estimated glomerular filtration rate (eGFR) < 80 mL/min, will be excluded.
12. Participants with severe cardiovascular or cerebrovascular disease, including unstable angina, heart failure classified as New York Heart Association (NYHA) class III or higher, or those in the acute phase of cerebral infarction, will be excluded.
13. Participants who are currently participating in another clinical trial will be excluded.
14. Participants with any other medical condition or circumstance that, in the opinion of the investigators, makes them unsuitable for participation will be excluded.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate of PCOS | Baseline and Week 24
  he proportion of participants who achieved regular menstrual cycles after 24 weeks of intervention and maintained regular cycles for at least 3 consecutive months.

SECONDARY OUTCOMES:
Waist circumference | Baseline, Week 12, and Week 24
Blood pressure | Baseline, Week 12, and Week 24
Weight | Baseline, Week 12, and Week 24
Body fat percentage | Baseline, Week 12, and Week 24
Skeletal muscle mass | Baseline, Week 12, and Week 24
Basal metabolic rate | Baseline, Week 12, and Week 24
Serum anti-Müllerian hormone (AMH) concentration | Baseline and Week 24
  Serum AMH levels will be measured in fasting serum samples collected at predefined study time points. Outcomes will be reported as circulating AMH concentrations and will be used to assess changes in ovarian reserve-related endocrine function between baseline and post-intervention time points and/or between intervention groups.
Progesterone | Baseline and Week 24
Fasting plasma glucose | Baseline and Week 24
Fasting insulin | Baseline and Week 24
Total cholesterol | Baseline and Week 24
Low-density lipoprotein cholesterol | Baseline and Week 24
High-density lipoprotein cholesterol | Baseline and Week 24
Triglycerides | Baseline and Week 24
Aspartate aminotransferase | Baseline and Week 24
Alanine aminotransferase | Baseline and Week 24
Dietary intake assessed by food frequency questionnaire (FFQ) | Baseline, Week 12, and Week 24
  Dietary intake will be assessed using a validated FFQ at predefined study time points. Outcomes will include quantitative estimates of habitual dietary intake, including energy and nutrient intakes, and comparisons of changes in dietary intake between study time points and/or between intervention groups.
Psychological status assessed by standardized questionnaire | Baseline, Week 12, and Week 24
  Psychological status will be assessed using a standardized, validated questionnaire administered at predefined study time points. Outcome measures will include questionnaire scores summarized as continuous variables, and changes in psychological status will be compared between baseline and post-intervention time points and/or between intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Gao, Doctoral degree, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and the need to protect sensitive participant information. Sharing the data could potentially breach confidentiality agreements and ethical guidelines, as the de-identified data might still be traceable back to participants. Additionally, the research team has not obtained prior consent for data sharing, and sharing IPD would require additional approvals from the ethics committee and participants.